CLINICAL TRIAL: NCT03950089
Title: Optical Coherence Tomography Angiography (OCT-A) Quantitative Assessment of Choriocapillaris Blood Flow in Central Serous Chorioretinopathy (CSC)
Brief Title: Optical Coherence Tomography Angiography (OCT-A) and Central Serous Chorioretinopathy (CSC)
Acronym: OPACITY
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: OCTA CSC
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Central Serous Chorioretinopathy
  Interventions: Device: Optical Coherence Tomography Angiography (OCT-A)
- Healthy patients
  Interventions: Device: Optical Coherence Tomography Angiography (OCT-A)

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography (OCT-A) — Optical Coherence Tomography Angiography (OCT-A) images were acquired using an Spectral Domain Optical Coherence Tomography device (Cirrus High Definition OCT Model 5000 with Angioplex; Carl Zeiss Meditec, Dublin, California, USA). With an acquisition speed of 68,000 A-Scan per second, the OCT Microangiography Complex algorithm provided OCT-A information for three-dimensional (3D) flow reconstruction. At each visit, each subject underwent a 3 x 3 millimeter (mm) macular 3D cube acquisition in both eyes. FastTrac continuous eye tracking technology was employed to control for eye movements and minimize motion artefacts.

SUMMARY:
Optical Coherence Tomography Angiography (OCT-A) is a noninvasive imaging technique that allows one to see blood vessels in the retina. The investigating team used this approach in patients with acute, recurrent and persistent subtypes of Central Serous Chorioretinopathy (CSC) to check for possible Choriocapillaris hypoperfusion. The presence or absence of these microvascular changes was explored in both eyes of the patients and compared to a control group of healthy volunteers. The possibility of a correlation between Choriocapillaris flow deficits, age and spontaneous resolution of serous retinal detachment was also evaluated. This study was conducted in an effort to improve one's understanding of this disease and other pachychoroid disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute, recurrent or persistent forms of central serous chorioretinopathy

Exclusion Criteria:

* Patients with chronic central serous chorioretinopathy were not eligible for inclusion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute, recurrent or persistent forms of central serous chorioretinopathy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Total number average individual area of flow signal voids | 2 months
  3x3 Optical Coherence Tomography Angiography (OCT-A) images on choriocapillaris slab were exported from the Angioplex software and then imported into the open-source Fiji software. Each image was binarized in black and white pixels. Thresholded areas greater than or equal to 1 white pixel were considered as flow signal voids
Total area of flow signal voids | 2 months
  3x3 Optical Coherence Tomography Angiography (OCT-A) images on choriocapillaris slab were exported from the Angioplex software and then imported into the open-source Fiji software. Each image was binarized in black and white pixels. Thresholded areas greater than or equal to 1 white pixel were considered as flow signal voids

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Mathis, MD, Principal Investigator — Hospices Civils de Lyon